CLINICAL TRIAL: NCT06419231
Title: A Double-blind, Randomized, Placebo-controlled Study to Evaluate the Effects of a Butyrate Formulation and a Butyrate + Polyphenol Formulation on Gut Health, Permeability and Associated Symptoms
Brief Title: Effectiveness of a Butyrate Formulation and Butyrate + Polyphenol Formulation on Gut Health, Permeability and Associated Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supplement Formulators, Inc. (Industry)
Collaborators: Compound Solutions Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL115
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Gut Health
Keywords: Gastrointestinal discomfort; Abdominal pain; Gas; Bloating; Diarrhea; Constipation; Heartburn; Abdominal discomfort
MeSH Terms: conditions — Abdominal Pain; Mucopolysaccharidosis IV; Diarrhea; Constipation; Heartburn | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Butyrate Formulation (Active Comparator): Butyrate Formulation: Take daily in the morning with 8 oz. (240ml) of water
  Interventions: Dietary Supplement: Butyrate Formulation
- Butyrate + Polyphenol Formulation (Active Comparator): Butyrate + Polyphenol Formulation: Take daily in the morning with 8 oz. (240ml) of water
  Interventions: Dietary Supplement: Butyrate + Polyphenol Formulation
- Placebo (Placebo Comparator): Placebo: Take daily in the morning with 8 oz. (240ml) of water
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Butyrate Formulation — Butyrate Formulation capsule: Take daily
  Arms: Butyrate Formulation
Dietary Supplement: Butyrate + Polyphenol Formulation — Butyrate + Polyphenol Formulation capsule: Take daily
  Arms: Butyrate + Polyphenol Formulation
Dietary Supplement: Placebo — Placebo: Take daily
  Arms: Placebo

SUMMARY:
The purpose of this study is the assess the effectiveness and safety of a Butyrate formulation and a Butyrate + Polyphenol formulation on gut health, permeability and associated symptoms

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled, remote design study to evaluate the effects of a Butyrate formulation and Butyrate + Polyphenol formulation on gut health, intestinal permeability and associated symptoms.

Participants will be asked to complete laboratory assessments and questionnaires. A total of up to 105 subjects (35 subjects per arm) will be enrolled in a randomly assigned sequence for the 28-day period. There will be scheduled remote video calls during the study.

The study subjects will complete assessment tools that include a Rating Scale for Gastrointestinal Symptoms, Quality of Life Questionnaire for Digestion, Visual Analogue Scale of Abdominal Pain, Stool Form Scale, Global Assessment of Improvement Scale-Gastrointestinal and the Short Form-36 Health Survey (SF-36). Laboratory testing will include an assessment of Gut Microbiome, analysis of Short Chain Fatty Acids, a panel for the Gut Barrier and Intestinal Permeability.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory, male or female, 21-70 years of age
2. A BMI of 18.5 -34.9
3. . Experiences at least three conditions involving gastrointestinal health on a weekly basis
4. Are comfortable fasting overnight
5. Are able to complete study procedures for up to approximately 6 hours on 2 separate days
6. Considered to be generally healthy on the basis of medical history
7. Willing to follow study instructions, including compliance with the study procedures and requirements

Exclusion Criteria:

1. Unable to provide a urine specimen, stool specimen or blood sample from a finger stick
2. Currently on a galactose/lactose restricted diet
3. Having taken proton pump inhibitors within the past 3 months
4. History of oral antibiotic use within the past 3 months
5. Current or previous history of gastrointestinal disease, cancer, infection or surgery that may interfere with the outcome parameters
6. A medical or surgical event requiring hospitalization, outpatient visits or emergency room visits within the past 5 years or in the judgment of the Study Investigator /Sub-I would preclude participation in the study
7. Current or previous history of diabetes
8. History of a major change in dietary habits with the past 1 month
9. Known intolerance or allergy to sugar alcohols including mannitol, sorbitol, xylitol, lactulose or lactose
10. Women who are lactating, pregnant or planning pregnancy within the next two months
11. Having donated blood or received a blood transfusion within 30 days before screening
12. Currently participating in another clinical research study or participated in another clinical research study within 30 days prior to screening

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-06-18 (Actual)

PRIMARY OUTCOMES:
Assessment of Gut Microbiome | 28 days
  Assessment of the median change in the results of the Gut Microbiome from baseline.
The Gastrointestinal Symptom Rating Scale (GSRS) Irritable Bowel Syndrome (IBS) version | 28 days
  Assessment of the median change in the responses on the Gastrointestinal Symptom Rating Scale-IBS from baseline. This scale has questions about how you have been feeling and what it has been like in the past week. The responses to each question range from no discomfort at all to very severe discomfort which would indicate a worse outcome.

SECONDARY OUTCOMES:
Gut Barrier Panel | 28 days
  Assessment of the median change in the results of the Panel for the Gut Barrier from baseline.
Short Chain Fatty Acids (SCFA) | 28 days
  Assessment of the median change in the results of the Short Chain Fatty Acid Analysis from baseline.
Intestinal Permeability Test | 28 days
  Assessment of the median change in the results of the Intestinal Permeability Test from baseline.
Digestion - Associated Quality of Life Questionnaire (DQLQ) | 28 days
  Assessment of the median change in the responses on the Digestion- Associated Quality of Life Questionnaire (DQLQ) from baseline. The questionnaire has questions related to digestive events and experiences in the last seven days evaluated on a scale from never (0%) to always (100%). The lower score indicates an improved outcome.
Visual Analogue Scale (VAS) of abdominal pain | 28 days
  Assessment of the median change in the responses on the Visual Analogue Scale questionnaire of abdominal pain from baseline. This scale indicates the response to the intensity of abdominal pain at the time evaluated on a scale from 0 (no pain) to 10 (severe pain). The lower the value indicates an improved outcome.
Bristol Stool Form Scale (English for United States) | 28 days
  Assessment of the median change in the stool form from baseline. This is related to asking the subject what their stool looked like each time they had a bowel movement for the day. There are 7 various stool types to choose ranging from Type 1 to Type 7. Types 3 or 4 are the preferred types.
Gastrointestinal- Global Assessment of Improvement Scale (Gastrointestinal-GAI) | 28 days
  Assessment of the median change in the responses on the Gastrointestinal- Global Assessment of Improvement Scale from baseline. This scale indicates the status of the gastrointestinal symptoms over the past 7 days. The responses range from substantially worse to substantially improved which would indicate an improved outcome.
Short Form-36 Health Survey (SF-36 Health Survey) | 28 days
  Assessment of the median change in the responses to the SF-36 Health Survey from baseline. This is a 36-item questionnaire that covers eight domains including physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue and general health perceptions. The scores from each domain can range from 0 to 100. The higher the scores for each domain indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Swick, Ph.D, Principal Investigator — Life Extension
Locations (1):
- Life Extension Clinical Research, Inc., Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asbaghi O, Nazarian B, Reiner Z, Amirani E, Kolahdooz F, Chamani M, Asemi Z. The effects of grape seed extract on glycemic control, serum lipoproteins, inflammation, and body weight: A systematic review and meta-analysis of randomized controlled trials. Phytother Res. 2020 Feb;34(2):239-253. doi: 10.1002/ptr.6518. Epub 2019 Dec 26. PMID 31880030
- [Background] Banasiewicz T, Krokowicz L, Stojcev Z, Kaczmarek BF, Kaczmarek E, Maik J, Marciniak R, Krokowicz P, Walkowiak J, Drews M. Microencapsulated sodium butyrate reduces the frequency of abdominal pain in patients with irritable bowel syndrome. Colorectal Dis. 2013 Feb;15(2):204-9. doi: 10.1111/j.1463-1318.2012.03152.x. PMID 22738315
- [Background] Brooker S, Martin S, Pearson A, Bagchi D, Earl J, Gothard L, Hall E, Porter L, Yarnold J. Double-blind, placebo-controlled, randomised phase II trial of IH636 grape seed proanthocyanidin extract (GSPE) in patients with radiation-induced breast induration. Radiother Oncol. 2006 Apr;79(1):45-51. doi: 10.1016/j.radonc.2006.02.008. Epub 2006 Mar 20. PMID 16546280
- [Background] Canani RB, Costanzo MD, Leone L, Pedata M, Meli R, Calignano A. Potential beneficial effects of butyrate in intestinal and extraintestinal diseases. World J Gastroenterol. 2011 Mar 28;17(12):1519-28. doi: 10.3748/wjg.v17.i12.1519. PMID 21472114
- [Background] Cleophas MCP, Ratter JM, Bekkering S, Quintin J, Schraa K, Stroes ES, Netea MG, Joosten LAB. Effects of oral butyrate supplementation on inflammatory potential of circulating peripheral blood mononuclear cells in healthy and obese males. Sci Rep. 2019 Jan 28;9(1):775. doi: 10.1038/s41598-018-37246-7. PMID 30692581
- [Background] Conley BA, Egorin MJ, Tait N, Rosen DM, Sausville EA, Dover G, Fram RJ, Van Echo DA. Phase I study of the orally administered butyrate prodrug, tributyrin, in patients with solid tumors. Clin Cancer Res. 1998 Mar;4(3):629-34. PMID 9533530
- [Background] Cory H, Passarelli S, Szeto J, Tamez M, Mattei J. The Role of Polyphenols in Human Health and Food Systems: A Mini-Review. Front Nutr. 2018 Sep 21;5:87. doi: 10.3389/fnut.2018.00087. eCollection 2018. PMID 30298133
- [Background] Costa C, Tsatsakis A, Mamoulakis C, Teodoro M, Briguglio G, Caruso E, Tsoukalas D, Margina D, Dardiotis E, Kouretas D, Fenga C. Current evidence on the effect of dietary polyphenols intake on chronic diseases. Food Chem Toxicol. 2017 Dec;110:286-299. doi: 10.1016/j.fct.2017.10.023. Epub 2017 Oct 14. PMID 29042289
- [Background] Dallal, G. (2021). www.Randomization.com. http://www.randomization.com
- [Background] Drugs, O. o. N. (2005). Guidance for Industry Estimating the Maximum Safe Starting Dose in Initial Clinical Trials for Therapeutics in Adult Healthy Volunteers. Office of the Federal Register National Archives and Record Administration
- [Background] Edelman MJ, Bauer K, Khanwani S, Tait N, Trepel J, Karp J, Nemieboka N, Chung EJ, Van Echo D. Clinical and pharmacologic study of tributyrin: an oral butyrate prodrug. Cancer Chemother Pharmacol. 2003 May;51(5):439-44. doi: 10.1007/s00280-003-0580-5. Epub 2003 Mar 12. PMID 12736763
- [Background] Grosicki, G. (2021). Effects of 3-week Tributyrin Supplementation on the Gut Microbiome: A Pilot Study. Journal of the Academy of Nutrition and Dietetics, 121(9, Supplement), A23. https://doi.org/https://doi.org/10.1016/j.jand.2021.06.051
- [Background] Hodges, J., Zeng, M., Cao, S., Pokala, A., Rezaei, S., Sasaki, G., Vodovotz, Y., & Bruno, R. (2022). Catechin-Rich Green Tea Extract Reduced Intestinal Inflammation and Fasting Glucose in Metabolic Syndrome and Healthy Adults: A Randomized, Controlled, Crossover Trial. Current Developments in Nutrition, 6(Supplement_1), 981-981. https://doi.org/10.1093/cdn/nzac068.010
- [Background] Hodgkinson K, El Abbar F, Dobranowski P, Manoogian J, Butcher J, Figeys D, Mack D, Stintzi A. Butyrate's role in human health and the current progress towards its clinical application to treat gastrointestinal disease. Clin Nutr. 2023 Feb;42(2):61-75. doi: 10.1016/j.clnu.2022.10.024. Epub 2022 Nov 2. PMID 36502573
- [Background] Istas G, Wood E, Le Sayec M, Rawlings C, Yoon J, Dandavate V, Cera D, Rampelli S, Costabile A, Fromentin E, Rodriguez-Mateos A. Effects of aronia berry (poly)phenols on vascular function and gut microbiota: a double-blind randomized controlled trial in adult men. Am J Clin Nutr. 2019 Aug 1;110(2):316-329. doi: 10.1093/ajcn/nqz075. PMID 31152545
- [Background] Kapolou, A., Karantonis, H. C., Rigopoulos, N., & Koutelidakis, A. E. (2021). Association of Mean Daily Polyphenols Intake with Mediterranean Diet Adherence and Anthropometric Indices in Healthy Greek Adults: A Retrospective Study. Applied Sciences, 11(10), 4664. https://www.mdpi.com/2076-3417/11/10/4664
- [Background] Le Sayec M, Xu Y, Laiola M, Gallego FA, Katsikioti D, Durbidge C, Kivisild U, Armes S, Lecomte M, Fanca-Berthon P, Fromentin E, Plaza Onate F, Cruickshank JK, Rodriguez-Mateos A. The effects of Aronia berry (poly)phenol supplementation on arterial function and the gut microbiome in middle aged men and women: Results from a randomized controlled trial. Clin Nutr. 2022 Nov;41(11):2549-2561. doi: 10.1016/j.clnu.2022.08.024. Epub 2022 Sep 6. PMID 36228567
- [Background] Ljotsson B, Jones M, Talley NJ, Kjellstrom L, Agreus L, Andreasson A. Discriminant and convergent validity of the GSRS-IBS symptom severity measure for irritable bowel syndrome: A population study. United European Gastroenterol J. 2020 Apr;8(3):284-292. doi: 10.1177/2050640619900577. Epub 2020 Jan 14. PMID 32213021
- [Background] Ma, G., & Chen, Y. (2020). Polyphenol supplementation benefits human health via gut microbiota: A systematic review via meta-analysis. Journal of Functional Foods, 66, 103829. https://doi.org/https://doi.org/10.1016/j.jff.2020.103829
- [Background] Park SY, Kim YD, Kim MS, Kim KT, Kim JY. Cinnamon (Cinnamomum cassia) water extract improves diarrhea symptoms by changing the gut environment: a randomized controlled trial. Food Funct. 2023 Feb 6;14(3):1520-1529. doi: 10.1039/d2fo01835g. PMID 36655542
- [Background] Pietrzak A, Banasiuk M, Szczepanik M, Borys-Iwanicka A, Pytrus T, Walkowiak J, Banaszkiewicz A. Sodium Butyrate Effectiveness in Children and Adolescents with Newly Diagnosed Inflammatory Bowel Diseases-Randomized Placebo-Controlled Multicenter Trial. Nutrients. 2022 Aug 11;14(16):3283. doi: 10.3390/nu14163283. PMID 36014789
- [Background] Recharla N, Geesala R, Shi XZ. Gut Microbial Metabolite Butyrate and Its Therapeutic Role in Inflammatory Bowel Disease: A Literature Review. Nutrients. 2023 May 11;15(10):2275. doi: 10.3390/nu15102275. PMID 37242159
- [Background] Rosner, B. (2006). Hypothesis Testing Two-Sample Inference. In Fundamentals of Biostatistics (6th ed., pp. 331-334). Duxbury Press.
- [Background] Wang X, Qi Y, Zheng H. Dietary Polyphenol, Gut Microbiota, and Health Benefits. Antioxidants (Basel). 2022 Jun 20;11(6):1212. doi: 10.3390/antiox11061212. PMID 35740109
- [Background] Zhang H, Liu S, Li L, Liu S, Liu S, Mi J, Tian G. The impact of grape seed extract treatment on blood pressure changes: A meta-analysis of 16 randomized controlled trials. Medicine (Baltimore). 2016 Aug;95(33):e4247. doi: 10.1097/MD.0000000000004247. PMID 27537554